CLINICAL TRIAL: NCT03981731
Title: Management of Perioperative Anxiety by the Fixed Rate Guided Breathing Technique (Cardiac Coherence) Coupled With a Hypnosis Session, as Part of the Improved Pre-habilitation After Surgery
Brief Title: Management of Perioperative Anxiety by the Cardiac Coherence Technique Coupled With a Hypnosis Session
Acronym: COHEC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut du Cancer de Montpellier - Val d'Aurelle (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: PROICM 2019-06 COH
Record Dates: First submitted 2019-06-07; First posted 2019-06-11 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Breast Cancer; Gynecologic Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cardiac coherence (Experimental)
  Interventions: Other: Cardiac coherence

INTERVENTIONS:
Other: Cardiac coherence — An initiation session to cardiac coherence will take place between D-10 and D-7 before the operation (during the anaesthesia consultation) in order to obtain a breathing rate of 6 cycles/min via a free application (Respirelax) with listening to an audio tape.
  3 cardiac coherence sessions per day of 5 min (before meals) during the 7 days preceding the operation.
  - The anaesthetic induction will be done with a session of cardiac coherence associated with listening to the audio tape.

SUMMARY:
the investigator proposes to use the cardiac coherence technique coupled with a hypnosis session to improve post-operative recovery.

DETAILED DESCRIPTION:
The perioperative period is recognized as an anxiety-provoking period for patients. If for some patients, this anxiety is more or less manageable, for others, it is the major concern with regard to their intervention, fearing not to wake up, to remain in a coma. Consideration of this aspect is very important for patients who require surgery. It is also a concern for caregivers involved in the care of these patients, including anesthesiologists, surgeons and operating room staff.

For many years, pharmacological premedication, including benzodiazepines, has been the gold standard in the treatment of preoperative anxiety.

This systematic prescription is controversial in populations most exposed to side effects such as the elderly, patients with heart or respiratory diseases.

Surgery also seems to influence the impact of premedication. For example, abdominal surgery and breast surgery are associated with a higher risk of agitation upon awakening.

Mental preparation, based on simple explanations by the anaesthetist, is not enough to reduce patients' anxiety.

A recent study evaluated the perioperative experience of patients receiving or not receiving premedication. It shows that benzodiazepines are associated with cognitive impairment and delayed extubation in the elderly. In addition, it seems to have little effect on patient anxiety when compared to a placebo.

In this context of anxiety, an emotional regulation tool appears particularly relevant. Cardiac coherence" (CC) is a particular state of cardiac variability. This state is correlated with many physiological and psychological variables. It is possible to promote this state through different techniques. One of its practices, "fixed frequency guided breathing", seems relevant both in its principles and in its simplicity of implementation.

This specific respiratory mode permits to rebalance the sympathetic - parasympathetic balance of the autonomic nervous system and reveals a state of calm vigilance. This simple, well-coded respiratory psychophysiological practice is widely used in many applications, such as for the most caricatural ones, the management of difficult situations where stress is a central element such as decision-making among fighter pilots on mission, in national education to improve academic learning (especially among anxious students) and also more generally in stress and anxiety management.

This technique induces a refocusing of emotions by regulating the SNA and therefore a better regulation of the hormones involved in the emotional cascade.

This practice has several advantages:

* it is psychophysiological (psychocorporeal) and widely described in the scientific literature in several indications
* it is completely free of charge and immediately accessible to the patient, regardless of time and place
* it can be used at other anxiety-inducing times (e.g., imaging or biopsy tests)
* it allows total patient autonomy, offering self-management of anxiety and independence from the presence of a third party
* it can approach a hypnotic model by focusing and absorbing what it can induce on breathing, and thus share some of its benefits
* It does not have any adverse effects. The major difficulty of this technique is the adherence and regularity of the practice. The optimal effect is dependent on regular training.

To improve this adherence, an audio tape will be put online, read in a hypnotic tone, which will aim to explain respiratory physiology, the benefits of oxygenation on cells and metabolism; this will have the effect of understanding the interest and utility of this exercise and will contribute to induce a feeling of relaxation and well-being.

This study will be a study of feasibility about a program based on the cardiac coherence technique in a context of perioperative anxiety.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years old
2. Surgery for breast or gynaecological cancer requiring scheduled hospitalization for up to 3 days
3. Signing of informed consent before any specific procedure in the study
4. Patient affiliated to a social security system

Exclusion Criteria:

1. Patients undergoing outpatient surgery for their cancer will not be included
2. Natural bradycardia (50 beats per minute)
3. Patient taking β-blockers, digoxin, flecaine, isoptin, cordarone, diltiazem
4. Cardiac arrhythmias
5. Severe heart failure with ventricular ejection fraction < 40%
6. Uncontrolled chronic pain
7. Patients whose medical or psychological conditions do not allow them to complete the study or sign the consent
8. Patient does not understand the French language
9. Deaf and/or dumb patient
10. Adult patient under guardianship or curatorship

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2020-02-14 (Actual); Primary Completion 2022-01-14 (Actual); Study Completion 2022-01-14 (Actual)

PRIMARY OUTCOMES:
Proportion of patients who have enrolled in the pre-habilitation program | 7 days
  A patient will be considered to have optimally adhered to the program if she performs at least 2/3 of the proposed cardiac coherence sessions (that represents 67% of the total number of sessions), that is, at least 14 sessions over the 7 days preceding the surgery.

SECONDARY OUTCOMES:
The preoperative anxiety score by using the Amsterdam Preoperative Anxiety and Information Scale (APAIS) | 7 days
  The anxiety scale consists of six items, each of which could be scored from 1 to 5 with the end poles "not at all" (1) and "extremely" (5). The score of the anxiety scale is the sum of these four questions, with a scoring range from 6 to 30.
Patient's satisfaction with perioperative period by using "Evaluation of the Vecu of General Anesthesia" questionnaire (EVAN-G) | 48 hours
  The validated EVAN-G questionnaire includes 26 questions whose results are grouped together to define 6 "dimensions": Attention Focus, Information, Privacy, Pain, Discomfort and Wait Times. From these scores, an overall satisfaction score is calculated (average of all scores). For each of the scores: the higher the score, the higher the satisfaction. For each dimension, scores were reduced on a scale from 0 to 100. The higher the score, the higher the perceived quality of the experience. The total score was the sum of the scores of the six dimensions reduced to 100.
Measurement of the Postoperative Quality of Recovery (QoR) | 10 days
  The quality of postoperative functional recovery will be assessed by the QoR-15 questionnaire, which assesses five dimensions of recovery (physical comfort ; emotional state ; physical independence ; physiological support ; and pain). Each item was rated on a ten-point Likert scale: none of the time, some of the time, usually, most of the time, and all the time. The total score on the QoR-15 ranges from 0 (poorest quality of recovery) to 150 (best quality of recovery).
Measurement of anxiety level by using a visual analogue scale | 7 days
  It's a visual scale from 0 (no anxiety) to 100 (highest anxiety)
Measurement of wake-up quality by using a visual analogue scale | 1 day
  It's a visual scale from 0 (best wake-up) to 100 (worst wake-up)
Measurement of post-operative pain by using a visual analogue scale | 1 day
  It's a visual scale from 0 (no pain) to 100 (highest pain)
Measurement of post-operative fatigue by using a visual analogue scale | 1 day
  It's a visual scale from 0 (no fatigue) to 100 (highest fatigue)
Measurement of comfort and satisfaction with care by using a visual analogue scale | 1 day
  It's a visual scale from 0 (ideal care) to 100 worst care)
Number of patients taking anesthetic drugs at induction of anaesthesia | 1 day
Number of patients taking anesthetic drugs during the post-interventional monitoring | 1 day
Number of patients taking morphine in recovery room | 1 day
Number of patients taking setrons (nausea and vomiting medication) | 1 day
Rate of patients that consider continuing the program of cardiac coherence | 1 day
Rate of patients willing to recommend the technique | 1 day
Number of days of hospitalization | 1 month
Number of patients taking morphine in peroperative | 1 day
Measurement of pain at inclusion by using a visual analogue scale | 1 day
  It's a visual scale from 0 (no pain) to 100 (highest pain)
The recruitment rate (proportion of patients consenting to participate in the study among eligible patients at the screening) and reasons for refusal. | 1 day

CONTACTS AND LOCATIONS:
Overall Officials: Jibba AMRAOUI, MD, Study Chair — Institut régional du cancer de Montpellier
Locations (1):
- Institut régional du cancer de Montpellier, Montpellier, Hérault, France

IPD SHARING:
Plan to Share IPD: Yes
All data will be available after publication of the results in peer-reviewed revues, and in national and international meetings. It includes all disidentified participants' data, the study protocol, the statistical analysis plan, the clinical study report and the analytic code. The corresponding author will provide data and datasets generated and/or analyzed during the study upon reasonable request.
Supporting Information: Study Protocol, SAP, CSR, Analytic Code
Time Frame: Access to study data upon written detailed request sent to ICM after publication.
Access Criteria: The data shared will be limited to that required for independent mandated verification of the published results, the applicant will need authorization from ICM for personal access, and data will only be transferred after signing of a data access agreement.

REFERENCES:
- [Background] Pekcan M, Celebioglu B, Demir B, Saricaoglu F, Hascelik G, Yukselen MA, Basgul E, Aypar U. The effect of premedication on preoperative anxiety. Middle East J Anaesthesiol. 2005 Jun;18(2):421-33. PMID 16438017
- [Background] Van den Bosch JE, Moons KG, Bonsel GJ, Kalkman CJ. Does measurement of preoperative anxiety have added value for predicting postoperative nausea and vomiting? Anesth Analg. 2005 May;100(5):1525-1532. doi: 10.1213/01.ANE.0000149325.20542.D4. PMID 15845719
- [Background] Munoz HR, Dagnino JA, Rufs JA, Bugedo GJ. Benzodiazepine premedication causes hypoxemia during spinal anesthesia in geriatric patients. Reg Anesth. 1992 May-Jun;17(3):139-42. PMID 1606095
- [Background] Agelink MW, Majewski TB, Andrich J, Mueck-Weymann M. Short-term effects of intravenous benzodiazepines on autonomic neurocardiac regulation in humans: a comparison between midazolam, diazepam, and lorazepam. Crit Care Med. 2002 May;30(5):997-1006. doi: 10.1097/00003246-200205000-00008. PMID 12006794
- [Background] Lepouse C, Lautner CA, Liu L, Gomis P, Leon A. Emergence delirium in adults in the post-anaesthesia care unit. Br J Anaesth. 2006 Jun;96(6):747-53. doi: 10.1093/bja/ael094. Epub 2006 May 2. PMID 16670111
- [Background] McCraty R, Atkinson M, Tiller WA, Rein G, Watkins AD. The effects of emotions on short-term power spectrum analysis of heart rate variability. Am J Cardiol. 1995 Nov 15;76(14):1089-93. doi: 10.1016/s0002-9149(99)80309-9. PMID 7484873
- [Result] Amraoui J, Leclerc G, Jarlier M, Diaz J, Guler R, Demoly C, Verin C, Rey Dit Guzer S, Chalbos P, Moussion A, Taoum C, Neron M, Philibert L. Cardiac coherence and medical hypnosis: a feasibility study of a new combined approach for managing preoperative anxiety in patients with breast or gynaecological cancer. BJA Open. 2024 Sep 24;12:100309. doi: 10.1016/j.bjao.2024.100309. eCollection 2024 Dec. PMID 39381542